CLINICAL TRIAL: NCT06611930
Title: A Randomized, Double-blind, Placebo-controlled Proof-of-concept Parallel Group Clinical Trial to Investigate the Efficacy, Safety and Tolerability of Weekly Subcutaneous Dosing of CK-0045 in Participants With Overweight/Obesity and Type 2 Diabetes
Brief Title: CK-0045 Proof-of-concept Study in Participants With Overweight / Obesity and Type 2 Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cytoki Pharma (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry); CRS Clinical Research Services Mannheim GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CK-0045_CS02
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Obesity and Overweight
Keywords: CK-0045
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Parallel group clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CK-0045 Dose level 1 (Experimental)
  Interventions: Drug: CK-0045
- CK-0045 Dose level 2 (Experimental)
  Interventions: Drug: CK-0045

INTERVENTIONS:
Drug: CK-0045 — Interleukin-22 agonist
  Arms: CK-0045 Dose level 1; CK-0045 Dose level 2
Drug: Placebo — Placebo (liquid for injection, which includes no active ingredient).
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if treatment with CK-0045 improves blood sugar control after a meal in participants with type 2 diabetes mellitus (T2DM) and overweight/obesity. It also aims to learn if CK-0045 can reduce body weight in these patients.

The main question it aims to answer is:

• Does 16 weeks of treatment with CK-0045 improve blood sugar control after a meal in participants with overweight or obesity and T2DM? Researchers will compare two dose levels of CK-0045 to a placebo arm (a look-alike substance that contains no drug) to see if CK-0045 improves blood sugar control.

Participants will:

* Have CK-0045 or placebo injected subcutaneously (under the skin) once weekly over a period of 16 weeks.
* Visit the clinic 24 times and stay overnight at 2 of the visits.
* During the visits blood samples will be collected and several other assessments/examinations will be performed to learn about the effects (and potential side effects) of CK-0045.

DETAILED DESCRIPTION:
Phase 2a, randomized, double-blind, placebo-controlled, parallel group trial with weekly SC dosing of CK-0045 (2 dose levels) or placebo over 16 weeks followed by 8 weeks of follow-up in participants with overweight / obesity and T2DM. The total duration of involvement for each participant, screening through follow-up, will be approximately 30 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* 18-74 years old male or female diagnosed with type 2 diabetes mellitus ≥ 6 months prior to screening
* Body Mass Index (BMI) between 27.0 and 40.0 kg/m^2 at screening
* Treated with diet and exercise
* HbA1c 6.5-8.5%, both inclusive, at screening for participants taking 3 antidiabetic medications or HbA1c 6.5-9.0%, both inclusive, at screening for participants taking 2 or less antidiabetic medications at stable doses for at least 3 months prior to screening

Key Exclusion Criteria:

* Any of the following within the past 6 months prior to screening: myocardial infarction, unstable angina, coronary artery bypass graft, percutaneous coronary intervention (diagnostic angiograms are permitted), transient ischemic attack, cerebrovascular accident or decompensated congestive heart failure, or currently have New York Health Association Class III or IV heart failure or any other clinically significant history or evidence of poorly controlled cardiovascular disorder(s) as judged by the investigator.
* Have a known clinically significant gastric emptying abnormality (for example, severe diabetic gastroparesis or gastric outlet obstruction), have undergone gastric bypass (bariatric) surgery or restrictive bariatric surgery (for example, gastric banding ), and/or device-based therapy for obesity, or have had device removal within the past 6 months.
* History or signs of clinically relevant skin diseases including but not limited to: psoriasis, atopic dermatitis, eczema, etc., as judged by the investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-11-18 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Area under the plasma glucose (PG) curve after a MMTT (AUCPG(0-4h)) | 16 weeks

SECONDARY OUTCOMES:
Change from baseline in body weight | 16 weeks
Change from baseline in total cholesterol, HDL-, LDL-cholesterol, triglycerides, free fatty acids (FFA), and Lp(a) | 16 weeks
Change from baseline in HbA1c | 16 weeks
Ctrough, observed | 168 hours
  Ctrough, observed (Trough serum concentration observed at the end of the dosing interval (several visits))
Incidence of adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (2):
- Germany (2):
  - CRS Clinical Reserach Services Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Profil Institut für Stoffwechselforschung GmbH, Neuss

IPD SHARING:
Plan to Share IPD: No